CLINICAL TRIAL: NCT04987281
Title: Resection of Pulmonary Lesions Aided by Robotic Bronchoscopy With Cone CT and INdocyanin Green (REPLACING) Study
Brief Title: Robotic Bronchoscopy With Cone CT and Indocyanine Green to Aid Removal of Lung Lesions in Patients With Stage I Non-small Cell Lung Cancer or Lung Metastases, REPLACING Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: 0 ACTUAL Enrollment must have Overall Recruitment
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2021-0243; NCI-2021-05983 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0243 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-06-26; First posted 2021-08-03 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2023-12

CONDITIONS: Lung Non-Small Cell Carcinoma; Metastatic Malignant Neoplasm in the Lung; Stage I Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Device feasibility (bronchoscopy, CT, indocyanine green) (Experimental): During standard of care surgical resection, patients undergo robotic bronchoscopy and CT. Patients also receive indocyanine green via injection.
  Interventions: Procedure: Computed Tomography; Drug: Indocyanine Green Solution; Device: Therapeutic Bronchoscopy

INTERVENTIONS:
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: Indocyanine Green Solution — Given via injection
  Other Names: IC-GREEN; ICG Solution
Device: Therapeutic Bronchoscopy — Undergo bronchoscopy using Ion robotic bronchoscope

SUMMARY:
This phase II trial studies the use of Ion robotic bronchoscope with a mobile computed tomography (CT) scanner to biopsy tumors and inject a fluorescent dye called indocyanine green to mark the tumor during surgery in patients with stage I non-small cell lung cancer or cancer that has spread to the lung (lung metastases). Sometimes small tumors or those that are not on the surface of the lung can be challenging to remove without making larger incisions. Injecting the dye, may help doctors see the tumor more easily, which may allow for smaller incisions and by being able to see the tumor, doctors may be better able to decide where to make the incisions in order to get all of the tumor out.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the feasibility of using the Ion Endoluminal Platform (IEP; Intuitive, Sunnyvale, California [CA]) with the Cios Spin - a mobile cone-beam C - (Siemens Medical Solutions, Malvern, Pennsylvania [PA], United States [US]) in the operating room setting.

OUTLINE:

During standard of care surgical resection, patients undergo robotic bronchoscopy and CT. Patients also receive indocyanine green via injection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Medically operable
* Undergoing pulmonary resection for either stage I non-small cell lung cancer (NSCLC) (undergoing segmentectomy) or metastatic disease to the lung
* Lesions < 2cm in longest diameter
* Lesions are located at least 1cm from the pleura

Exclusion Criteria:

* Pregnant
* Serum creatinine > 2.0
* Central lesions
* Iodide allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Number of successful procedures out of 50 | through study completion, an average of 1 year
  Success is defined as the ability of the provider to navigate to the lesion and deploy the needle into the lesion using the three allotted scans to aid in targeting to the lesion (As evaluated by surgeon using cone beam computed tomography [CT]).

SECONDARY OUTCOMES:
Number of repositions required to deploy needle into lesion | through study completion, an average of 1 year
Presence or absence of diagnostic tissue in sample | Up to 2 years
  Evaluated using rapid cytology.
Indocyanine green visualized during robotic pulmonary resection | through study completion, an average of 1 year
Number of cases that were begun as robotic or video-assisted that were converted to open in order to palpate nodule | through study completion, an average of 1 year
Closest margin on resected nodule pathology | Up to 2 years
Proximity of needle to the lesion on first deployment | through study completion, an average of 1 year
  Evaluated retrospectively by research fellow using cone beam CT images.

CONTACTS AND LOCATIONS:
Overall Officials: David W Rice, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT04987281/ICF_000.pdf